CLINICAL TRIAL: NCT06265220
Title: A Phase 1 Study to Evaluate the Efficacy and Safety of AB-101, an Allogeneic Cord Blood- Derived NK-Cell Therapy in Combination With B-Cell Depleting mAb in Patients Who Failed Treatment for Class III or IV Lupus Nephritis or Other Forms of Refractory Systemic Lupus Erythematosus
Brief Title: AB-101 in Combination With B-Cell Depleting mAb in Patients Who Failed Treatment for Class III or IV Lupus Nephritis or Other Forms of Refractory Systemic Lupus Erythematosus
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Artiva Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AB-101-03
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Lupus Nephritis - WHO Class III; Lupus Nephritis - WHO Class IV; Refractory Systemic Lupus Erythematosus; SLE
Keywords: SLE; Lupus; Lupus Nephritis; AlloNK
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Cyclophosphamide; fludarabine; Rituximab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1: Dose confirmation of AB-101 as Monotherapy (Experimental)
  Interventions: Drug: AB-101; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 1: Dose confirmation of AB-101 plus Obinutuzumab combination (Experimental)
  Interventions: Drug: AB-101; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Obinutuzumab
- Phase 1: Dose confirmation of AB-101 plus Rituximab combination (Experimental)
  Interventions: Drug: AB-101; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab

INTERVENTIONS:
Drug: AB-101 — NK Cell Therapy
Drug: Cyclophosphamide — Lymphodepleting chemotherapy
Drug: Fludarabine — Lymphodepleting chemotherapy
Drug: Rituximab — Anti-CD20 antibody therapy
  Arms: Phase 1: Dose confirmation of AB-101 plus Rituximab combination
Drug: Obinutuzumab — Anti-CD20 antibody therapy
  Arms: Phase 1: Dose confirmation of AB-101 plus Obinutuzumab combination

SUMMARY:
AB-101 (also known as AlloNK) is an off-the shelf, allogeneic cell product made of "natural killer" cells, also called NK cells. White blood cells are part of the immune system and NK cells are a type of white blood cell that is known to enhance the effect of monoclonal antibody therapies.

This clinical trial will enroll adult patients with lupus nephritis Class III or IV either with or without the presence of Class V who relapsed or did not respond to previous standard of care treatment approaches, or other forms of refractory systemic lupus erythematosus.

The primary objective is to assess the safety, tolerability and preliminary activity of AB-101 plus a B-cell depleting mAb (e.g., rituximab, obinutuzumab) after cyclophosphamide and fludarabine in adult subjects with relapsed/refractory lupus nephritis Class III or IV, with or without the presence of Class V, or other forms of refractory systemic lupus erythematosus.

Patients will be assigned to receive either AB-101 alone as monotherapy or in combination with a B-cell depleting mAb (e.g., rituximab, obinutuzumab). All patients will receive at least 1 treatment cycle of AB-101, followed by scheduled assessments of overall health and response status.

Patients may receive up to 2 cycles of treatment spaced 24 weeks apart.

ELIGIBILITY:
Inclusion Criteria for all subjects (Lupus Nephritis or SLE)

* Diagnosis of SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) Classification Criteria
* Subjects must have had an inadequate response with at least two prior lines of standard of care (SoC) treatment.

Inclusion Criteria for LN:

* Adult subjects with lupus nephritis Class III or IV (with or without the presence of Class V)
* Evidence of active disease on renal biopsy.
* All subjects are required to receive adequate concomitant antihypertensive and antiproteinuric therapy with blockade of the renin-angiotensin system

Inclusion Criteria for SLE:

* Total systemic lupus erythematosus disease activity index (SLEDAI-2K score) ≥ 8, and clinical SLEDAI-2K ≥ 4.
* British Isles Lupus Assessment Group 2004 (BILAG-2004) activity score of A in ≥ 1 organ, or a BILAG-2004 activity score of B in ≥ 2 organs.
* Subjects have failed at least two conventional therapies

Exclusion Criteria:

* Known past or current malignancy
* Clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to SLE
* Subjects with known active viral infections
* Severe active CNS Lupus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events | From the time of consent through 104 weeks after initiation of study treatment
  Incidence, severity and causality of adverse events and serious adverse events
AB-101 Clinical Activity | From the time of first dose through 104 weeks after initiation of study treatment
  Determined by Overall Response Rate in subjects with lupus nephritis and refractory systemic lupus erythematosus

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saddekni, M.D., PgDip, BCMAS, Study Director — Artiva Biotherapeutics
Locations (9):
- United States (9):
  - Artiva Investigational Site Birmingham, Birmingham, Alabama
  - Artiva Investigational Site Tucson, Tucson, Arizona
  - Artiva Investigational Site San Diego, San Diego, California
  - Artiva Investigational Site Aventura, Aventura, Florida
  - Artiva Investigational Site Plantation, Plantation, Florida
  - Artiva Investigational Site Iowa, Iowa City, Iowa
  - Artiva Investigational Site Charlotte, Charlotte, North Carolina
  - Artiva Investigational Site Mesquite, Mesquite, Texas
  - Artiva Investigational Site Woodlands, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No
AlloNK is early in clinical development, next steps will be based on the progress of our data.